

**Statistical Analysis Plan** 

Phase I clinical study to evaluate the safety and tolerability of PRO-172 ophthalmic solution, manufactured by Laboratorios Sophia, SA de CV, on the ocular surface of ophthalmologically and clinically healthy subjects.



Creation date: September 2019.

Phase I clinical study to evaluate the safety and tolerability of PRO-172 ophthalmic solution, manufactured by Laboratorios Sophia, SA de CV, on the ocular surface of ophthalmologically and clinically healthy subjects.

Protocol Code: SOPH172-0919/I

Protocol Version: 0.1

#### Content

| 1.0 Abbreviations | 4 |
|----------------------------------------------|----|
| 2.0 Objectives of Study | 4 |
| 3.0 Hypothesis of Study | 5 |
| 4.0 Study Design | 5 |
| 4.1 Duration of treatment | 5 |
| Table 1. Study schedule | 5 |
| Figure 1. Study diagram | 8 |
| 5.0 Sample Size | 8 |
| 5.1 Sample Size Calculation | 8 |
| Statistical | 9 |
| 6.1 Primary outcome variables: | 9 |
| 6.2 Secondary outcome variables: | |
| Table 3. Operational Definition of Variables | 10 |
| 7.0 Methods of Analysis | 12 |
| Table 3. Triangulation of concepts | 14 |
| 8.0 Changes | 14 |
| 8.1 Author of the document: | 15 |

# Statistical Analysis Plan SOPH172-0919/I

## Bepostatin besylate 1.5%

| 9. | .0 References | .15 |
|-----|---------------------------------------------|-----|
| 7 ( | 0.0 Annexes | .16 |
| | 10.1 Eye comfort index | .16 |
| | 10.2 Efron scale for conjunctival hyperemia | .18 |
| | 10.3 Oxford Scale | .18 |

#### 1.0 Abbreviations

FCI Informed Consent Form

CRF Electronic Case Report Form

EA Adverse events

HC Conjunctival hyperemia

ITT Intention-to-treat population

LLS Safety call

MAVC Best corrected visual acuity

MC Concomitant medication

ICO Eye comfort index

PI Research Product

PIO Intraocular pressure

PP Population by protocol

PRO-172 Bepostatin besylate 1.5%

TRL Tear break-up time

VB Initial visit

VF Final visit

# 2.0 Objectives of the Study

To evaluate the safety and tolerability of the PRO-172 formulation manufactured by Laboratorios Sophia., SA de CV on the ocular surface of clinically healthy subjects.

## 3.0 Study Hypothesis

H $_{0}$ : PRO-172 ophthalmic solution is safe and tolerable in its ophthalmic application, presenting in less than 10% of the study population unexpected adverse events related to the investigational product.

H<sub>1</sub>: PRO-172 ophthalmic solution is not safe and tolerable for ophthalmic application, as it presented unexpected adverse events related to the investigational product in less than 10% of the study population.

## 4.0 Design of Study SOPH176-1218/I-II

Phase I clinical trial, controlled, non-comparative, open, single-center.

#### 4.1 Duration of treatment

7 days

Table 1. Study schedule.

| Procedures | VB | VF | LIS |
|-----------------------------|----|-----------|----------|
| Flocedules | DI | D 8 TO +1 | D 10 ± 1 |
| FCI SIGNATURE | Х | | |
| MEDICAL RECORD | Χ | | |
| CONCOMITANT MEDICATION | X | X | |
| EVALUATION | | ^ | |
| URINE PREGNANCY TEST | X | X | |
| VITAL SIGNS | X | X | |
| AVCC | X | X | |
| OCULAR SURFACE INTEGRITY | | | |
| (STAINING AND EVALUATION OF | Х | X | |
| CONJUNCTIVAL HYPEREMIA | | | |
| AND CHEMOSIS) | | | |

## Bepostatin besylate 1.5%

| COMPREHENSIVE | | | |
|------------------------------|---|---|---|
| OPHTHALMOLOGICAL | Χ | X | |
| EVALUATION | | | |
| PIO | X | Х | |
| ELIGIBILITY CRITERIA | Х | | |
| EA ASSESSMENT | Χ | Χ | X |
| RESEARCH PRODUCT (RP) | X | | |
| ASSIGNMENT | | | |
| EYE COMFORT INDEX | X | X | |
| DELIVERY OF THE PI AND START | X | | |
| OF INTERVENTION | ^ | | |
| DELIVERY OF THE SUBJECT'S | X | | |
| DIARY | ^ | | |
| ADHERENCE ASSESSMENT | | Х | |
| RETURN/EVALUATION OF THE | | Х | |
| SUBJECT'S DIARY | | ^ | |
| RETURN OF PI | | X | |



Figure 1. Study diagram.

### 5.0 Sample Size

A total size of 22 subjects is estimated, who will provide both eyes for the analysis.

### 5.1 Sample Size Calculation

Although there are no references on sample calculation in phase I studies, it was considered pertinent to do so according to the presence of Adverse Events (AE) reported by Macejko et al., 2010 [1], in a multicenter, double-blind, randomized, parallel-group controlled clinical trial. Where the efficacy and tolerability of a 1.5% bepotastine besilate ophthalmic solution (n=43) versus 1.0% bepotastine (n=44) and placebo (n=43) were evaluated in 130 subjects in a conjunctival allergen challenge (CARC) model.

The intervention consisted of the application of 3 drops in each eye of each of the interventions (3 minutes after the RAC), with measurements at 15 minutes, 8 and 16 hours post-instillation.

The percentage of adverse events was 30% for the 1.5% bepostatin group, 47.5% for 1% bepostatin, and 22.5% for placebo, so a non-inferiority margin of 10% was considered with the formulation proposed in this protocol (1.5% bepostatin) [1].

The sample size was calculated using the equation for a proportion [2], considering a power of 80% (  $\beta$  ), a significance level of 0.05 (  $\alpha$  ) and a non-inferiority margin (  $\delta$  ) of 10%.

Hypothesis

$$H_0: p - p_0 \leq \delta$$

$$H_1: p - p_0 > \delta$$

Where,  $\delta$  is the non-inferiority margin (-10%).

Equation

Bepostatin besylate 1.5%

The calculation to estimate the sample size and power was performed using the following equations.

$$n = p(1-p) \left( \frac{z_{1-\alpha} + z_{1-\beta}}{p - p_0 - \delta} \right)^2$$

$$1 - \beta = \theta(z - z_{1-\alpha}) + \theta(-z - z_{1-\alpha}), z = \frac{p - p_0 - \delta}{\sqrt{\frac{p(1-p)}{n}}}$$

Where:

n is the sample size,

pois the reference proportion,

 $\theta$  is the normal distribution function.

 $\alpha$  is the Type I error

 $\beta$  is the Type II error, which means that, 1-  $\beta$  is the power, and

 $\delta$  is the test margin.

Calculated sample: According to the previous calculation, the result is 18 subjects; this calculation was increased by 20% to account for possible losses. The total required sample size is 22 subjects, who will provide an input for the analysis.

## 6.0 Statistical Analysis Plan [3]

### 6.1 Primary outcome variables:

- Incidence of unexpected AEs related to the investigational product.
- ICO score.

### 6.2 Secondary outcome variables:

- Changes in Corrected Visual Acuity (CCVA).
- Corneal and conjunctival staining changes with lissamine green.
- Corneal and conjunctival staining changes with fluorescein.
- Changes in conjunctival hyperemia.
- Incidence of chemosis.

Table 3. Operational Definition of the Variables

| Variable | Conceptual<br>Definition | Operational<br>Definition | Type of measurement | Normal value | Statistical<br>test |
|---|---|---|---|---|---|
| Adverse<br>events | Any adverse medical event that occurs in a patient or clinical research subject who has been administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. [4] | Adverse events occurring during the study will be collected using the electronic CRF. | <ul> <li>Continuous quantitative.</li> <li>Qualitative categorical.</li> </ul> | <ul> <li>Frequency:</li> <li>Subjects presenting AE/Total number of exposed subjects.</li> <li>Intensity:</li> <li>O= Mild</li> <li>1= Moderate</li> <li>2= Severe</li> <li>Causality:</li> <li>O=Probably or possibly related.</li> <li>1=Unlikely related.</li> </ul> | • X <sup>2</sup> or<br>Fisher's<br>Exacta. |
| Ocular<br>Comfort<br>Index (OCI)<br>score. | The OIQ is a questionnaire designed to measure ocular surface irritation. It assesses symptoms focused on comfort associated with ocular surface disorders. Higher values indicate more severe symptoms. | The evaluator will administer the questionnaire to the subject and allow him or her to answer it calmly without any pressure or coercion. See Appendix 10.1, ICO. | Discrete<br>quantitative. | Score:<br>0=None,<br>100=High<br>discomfort. | • Wilcoxon rank test. |
| Changes in visual ability. | Best-corrected visual acuity (BCVA) is a test of visual function. Spatial VA is the ability to distinguish separate | Snellen chart | Discrete<br>quantitative. | Fraction,<br>normal value =<br>0.6 to 2.0 | • Wilcoxon rank test. |

| | | | | <u>Depostatiii De</u> | csylate 1.57 |
|---|---|---|---|---|---|
| | elements of an object and identify them as a whole. It is quantified as the minimum angle of separation (located at the nodal point of the eye) between two objects that allows them to be perceived as separate objects. | | | | |
| Corneal and conjunctival staining changes with lissamine green. | Detection of<br>epithelial defects in<br>the conjunctiva and<br>cornea. | Direct<br>observation with<br>a slit lamp,<br>Oxford scale<br>graduation. See<br>Appendix 10.3,<br>Oxford Scale. | Qualitative<br>Ordinal | Degrees: The staining is presented in a series of panels (AE). The staining points range from 0-5 for each panel and from 0-15 for the total exposed area of conjunctiva and cornea. | • X <sup>2</sup> or<br>Fisher's<br>Exacta. |
| Corneal and conjunctival staining changes with fluorescein. | Detection of<br>epithelial defects in<br>the conjunctiva and<br>cornea. | Direct observation with a slit lamp and cobalt blue filter, Oxford scale graduation. See Appendix 10.3, Oxford Scale. | Qualitative<br>Ordinal | Degrees: The staining is presented in a series of panels (AE). The staining points range from 0-5 for each panel and from 0-15 for the total exposed area of conjunctiva and cornea. | • X <sup>2</sup> or<br>Fisher's<br>Exacta. |

| Conjunctival<br>hyperemia<br>changes. | It is defined as the simplest reaction of the conjunctiva to a stimulus; a red appearance is observed secondary to vasodilation of the vessels of the conjunctiva of variable intensity. | Direct observation. Classification using the Efron scale. See Appendix 10.2, Efron Scale for Conjunctival Hyperemia. | Ordinal<br>qualitative. | Degrees: 0=Normal, 1= Very mild, 2= Mild, 3= Moderate, 4= Severe. | • X <sup>2</sup> or<br>Fisher's<br>Exacta. |
|---|---|---|---|---|---|
| Incidence of<br>Chemosis. | It is defined as conjunctival edema resulting from an inflammatory reaction. It is classified as present or absent. | The evaluator will use a narrow beam of light at 60° and measure whether the conjunctiva separates from the sclera by ≥1/3 of the total eyelid opening or if it extends beyond the gray line. | Qualitative<br>categorical. | 0=Absent<br>1= Present | • X <sup>2</sup> or<br>Fisher's<br>Exacta. |

# 7.0 Methods of Analysis [5]

Statistical analysis will be performed by personnel from Laboratorios Sophia, SA de CV. SPSS version 19.0 (IBM Corporation, Armonk, NY, USA) will be used. Coding will be performed using consecutive numbers. Data will be collected and organized in an Excel spreadsheet (Microsoft® Office). The data will then be exported to the SPSS platform. Variables will be categorized according to their nature (see Table 2).

Study participants will be identified by a number and their initials.

The initials of the subject of study will be obtained starting with the first letter of the name, followed by the first letter of the first surname and the first letter of the second surname, obtaining a maximum of three letters. In case the person has two names or a compound surname, the first letter will always be used.

### Example:

A. A rieh Daniel M ercado C arrizalez B. J uan D e la Torre O rozco

a. Initials: AMC b. Initials: JDO

Once the subject has been selected, they will be assigned a number that will identify them throughout the study. This code will consist of eight numbers in the following order from left to right:

- three digits of the molecule under study according to the name given by the sponsor.
- two digits corresponding to the research center number.
- three digits of the consecutive number assigned to its inclusion in the research center.

The Kolmogorov-Smirnov test will be performed to determine the distribution of the results obtained. [3]

The results of continuous quantitative variables will be presented in measures of central tendency: mean, standard deviation and ranges.

The statistical analysis of continuous quantitative variables to find significant differences ( p ) will be as follows:

• <u>Intra-group analysis:</u> They will be determined using the Wilcoxon rank test for quantitative variables. [6]

The level of difference to consider significance will be an alpha (  $\alpha$  ) of 0.05 or less.

The results of the nominal and ordinal qualitative variables will be presented in frequencies, proportions and percentages.

Statistical analysis to identify significant differences in qualitative variables will be performed by creating 2x2 contingency tables and will be carried out as follows:

• <u>Intra-group analysis: Pearson's Chi-square (X <sup>2</sup>) test or Fisher's exact test for expected values less than 5.</u>

The level of difference to consider significance will be an alpha (  $\alpha$  ) of 0.05 or less.

For adverse event reporting, all eyes of participants assigned to the intervention after the baseline visit will be considered. Results will be expressed as a percentage of subjects.

The final results report will be displayed in tables or graphs, as appropriate.

Table 3. Triangulation of concepts [5]

| Variable type | Variable | | В1 | B2 | C1 | C2 | DI | D2 | D3 | D4 |
|---|---|---|---|---|---|---|---|---|---|---|
| Background | | | | | | | | | | |
| A1 | Demographics | DT | | | | | | | | |
| Basal | | | | | | | | | | |
| B1 | Medical record | DT | | | | | | | | |
| B2 | DT | | | ТВ | | | | В | | |
| Security | | | | | | | | | | |
| C1 | EAs | | | | ТВ | В | В | TB | ТВ | ТВ |
| C2 | ICO | DB | | | В | В | | | | |
| Secondary outco | ome | | | | | | | | | |
| D1 | MAVC | DB | | | В | | В | | | |
| D2 | Ocular surface stains (TF and TVL). | DT | | | Т | | | Т | | |
| D3 | Conjunctival hyperemia | TD | | DT | Т | | | | Т | |
| D4 | Chemosis | TD | | DT | Т | | | | | Т |
| D, Descriptive statistics; T, 2x2 contingency table; B, Bivariate analysis; M, Multivariate analysis. | | | | | | | | | | |

## 8.0 Changes

Newly created document, no changes apply.

### 8.1 Author of the document:



#### 9.0 References

- 1. Macejko TT, Bergmann MT, Williams JKI., et al. Multicenter clinical evaluation of bepostatine besilate ophthalmic solutions 1.0% and 1.5% to treat allergic conjunctivitis. Am J Ophthalmol, 2010. 150(1): 122-7.
- 2. Chow S, Shao J, Wang H. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series, 2008: Chapter 4: 85-6.
- 3. Haffajee A., Socransky S. and Lindhe J. Comparison of statistical methods of analysis of data from clinical periodontal trials. *J Clin Periodontol*, 1983; 10: 247-256.
- 4. Mexican Official Standard NOM-220-SSA1-2016, Pharmacovigilance facilities and operations.
- 5. ICH E2A. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonized Tripartite Guideline. Clinical safety data management: definitions and standards for expedited reporting. October 1994.
- 6. Woolson R. Wilcoxon signed-rank test. *Wiley Encuclopedia of Clinical Trials, 2008,* pp. 1-3.

## 10.0 Annexes

# 10.1 Eye comfort index

| 11 000 00 | *********** | *********** | ************ | | ********** | | | *************************************** |
|---|---|---|---|---|---|---|---|---|
| Identification of | | | | | | _ | | |
| Study No.: SOPH172-0919-I | | | | | | | ate: / | ı |
| Subject's initia | ls: | | | | | Subject I | No.: 172 | |
| Directions: | | | | | | | | |
| This questionna | iro was do | signed to rat | e the comfo | d of your eyes | | | | |
| or each questi | | | e are conno | it or your eyes | | | | |
| Example: | | t week, how | often were y | our eyes red? | ' | | | |
| | Never<br>0 | 1 | 2 | 3 | 4 | 5 | Always | |
| here are no rig | iht or wrong | g answers. D | on't spend t | too much time | on each | question. | | |
| 4 | | | | | | | | |
| | ast week, h | now often die | your eyes | reel dry ? | | | | |
| <u>Never</u><br>0 | | 1 | 2 | 3 | | 4 | 5 | Always<br>6 |
| | | | - | | | , | | |
| When | our eves fe | It day how s | evere was t | he sensation ( | isually? | | | |
| I haven't fel | - | nt dry, now s | evere was t | ne sensauon u | isually: | | | Severe |
| 0 | C.R. | 1 | 2 | 3 | | 4 | 5 | 6 |
| 2 In the p | ast week. h | now often die | d vour eves t | feel aritty ? | | | | |
| Never | | | ., | y . | | | | Alwaye |
| 0 | | 1 | 2 | 3 | | 4 | 5 | Always<br>6 |
| When y | our eves fe | elt <i>aritty</i> , typic | cally, how in | tense was the | sensatio | on? | | |
| I haven't fel | | 3 3, 3, | ,. | | | | | Severe |
| 0 | | 1 | 2 | 3 | | 4 | 5 | 6 |
| 3 In the p | ast week, h | now often die | d your eyes t | feel throbbing | ? | | | |
| Never | | | | _ | | | | Always |
| 0 | | 1 | 2 | 3 | | 4 | 5 | 6 |
| When y | our eyes fe | elt like <i>they</i> w | vere stinging | , how intense | was the | sensation us | ually? | |
| I haven't fel | t it | | | | | | | Severe |
| 0 | | 1 | 2 | 3 | | 4 | 5 | 6 |
| 4 In the past v | veek, how o | often did you | ir eyes feel t | ired ? | | | | |
| Never | | | | | | | | Always |
| 0 | | 1 | 2 | 3 | | 4 | 5 | 6 |
| - | - | elt tired, how | intense was | the feeling us | sually? | | | |
| I haven't fel | t it | | | | | | | Severe |
| 0 | | 1 | 2 | 3 | | 4 | 5 | 6 |
| | | | | | | | | Sheet 1 of 2 |

# Statistical Analysis Plan SOPH172-0919/I

Bepostatin besylate 1.5%

| | | | | | Eye | comfort in | dex |
|---|---|---|---|---|---|---|---|
| 5 | In the past w | eek, how often | did your eyes fee | l sore ? | | | 1 |
| | Never | | | | | | Always_ |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | | | | | | | 1 |
| | When your ey | yes felt sore, h | ow severe was the | e sensation usu | ally? | | |
| - 1 | haven't felt it | | | | | | Severe |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | | | | | | | į |
| 6 | In the past w | eek, how often | did your eyes fee | l itchy? | | | |
| | Never | | | | | | Always_ |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | | | | | | | į |
| | When your ey | yes felt itchy , | how intense was t | he sensation us | ually? | | 1 |
| 1 | haven't felt it | | | | | | Severe |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |

 ${\it Ocular Comfort\ Index, translated\ from\ the\ Ocular\ Comfort\ Index\ available\ at:\ http://iovs.arvohournals.org}$ 

Sheet 2 of 2

# 10.2 Efron scale for conjunctival hyperemia



## 10.3 Oxford Scale

| PANEL | Grade | Criteria |
|-------|-------|-----------------------------------------------|
| A | 0 | Equal to or less than panel A |
| B | I | Equal to or less than panel B, greater than A |
| C | II | Equal to or less than panel C, greater than B |
| D | III | Equal to or less than panel D, greater than C |
| E | IV | Equal to or less than panel E, greater than D |
| >E | V | Greater than panel E |